CLINICAL TRIAL: NCT03133325
Title: A Randomized, Split Arm Study to Evaluate the Safety Following Injection of GP0045 Compared to Restylane Lyft Lidocaine
Brief Title: A Study to Evaluate the Safety Following Injection of GP0045 Compared to Restylane Lyft Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 43FE1629
Record Dates: First submitted 2017-04-18; First posted 2017-04-28 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2017-08

CONDITIONS: Safety
Keywords: Hyaluronic Acid, Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All subjects (Other): Treatment with both GP0045 and Restylane Lyft Lidocaine
  Interventions: Device: GP0045; Device: Restylane Lyft Lidocaine

INTERVENTIONS:
Device: GP0045 — Hyaluronic acid gel
Device: Restylane Lyft Lidocaine — Hyaluronic acid gel

SUMMARY:
This is a study to assess the safety of GP0045 compared to Restylane Lyft Lidocaine.

There is a 12-week follow-up period. AEs will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to adequately understand the verbal explanations and the written subject information provided in local language and ability to give consent to participate in the study
* Signed and dated informed consent to participate in the study, including photo consent
* Men or non-pregnant, non-breast feeding women aged 18 years or older

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any injectable HA gel
* Known/previous allergy or hypersensitivity to local anesthetics, e.g. lidocaine or other amide-type anesthetics
* Any condition (medical or other) that, in the opinion of the Investigator, would make the subject unsuitable for inclusion (e.g. a chronic, relapsing or hereditary disease that may interfere with the outcome of the study)
* Participation in any other clinical study within 30 days before treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the incidence, intensity, duration and onset of adverse events following injection of GP0045 | 12 weeks
  Incidence, intensity, duration, and onset of adverse events collected and assessed by the Investigator 12 weeks post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CTC, Uppsala, Sweden